CLINICAL TRIAL: NCT02190240
Title: Effect of Complementary and Alternative Medicine on Pain Among Inpatients
Status: Completed | Type: Observational
Sponsor: Allina Health System (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: AT006518-01; R01AT006518-01 (NIH)
Record Dates: First submitted 2014-07-08; First posted 2014-07-15 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Pain
Keywords: Complementary and Alternative Medicine; Integrative Medicine; Pain Management
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The proposed study has 3 aims: 1) quantitatively describe a model for delivering complementary and alternative medicine (CAM) therapies to understand the selection of patients and CAM therapies used for pain management, 2) examine the effects of selected CAM therapies on immediate change in pain, and 3) examine the effects of selected CAM therapies on duration of pain change.

Positive results from this study will assist hospitals in the integration of usual care and CAM therapy for pain reduction. Findings may also drive future research on the cost effectiveness of these therapies for pain management, as well as the impact on patient outcomes such as length of stay and use of narcotics.

ELIGIBILITY:
Aims 1 and 2 Inclusion Criteria:

* Admission to Abbott Northwestern Hospital
* Consent to release of electronic health record for research purposes
* 18 years of age or older
* Length of stay greater than 24 hours

Aims 1 and 2 Exclusion Criteria:

* None

Aim 3 Inclusion Criteria:

* Admission to Abbott Northwestern Hospital
* Length of stay greater than 24 hours
* 18 years of age or older
* Consent to release of electronic health record for research purposes
* Received CAM therapy in current hospitalization
* Pain level of 1 or greater at the pre-treatment assessment by practitioner
* English-speaking
* Integrative medicine therapy ended between 9:00 am and 4:00 pm

Aim 3 Exclusion Criteria:

* Refuses consent
* Unable to provide consent due to competency concerns
* Has declined study participation 3 times during current hospitalization
* Has hard declined during current hospitalization
* Has been approached 6 times during current hospitalization
* Has been approached to consent earlier that day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Abbott Northwestern Hospital Inpatients
Sampling Method: Non-Probability Sample
Enrollment: 4422 (Actual)
Dates: Start 2012-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Model of delivering CAM therapies | Up to 4 years
  Quantitatively describe a model for delivering CAM therapies to understand selection of patients and CAM therapies used for pain management.
Effects of selected CAM therapies on immediate change in pain | CAM Visit (30-45 minutes)
  We will examine the effectiveness of CAM therapies on self-reported (11 point scale) pain measured just before and immediately after service delivery.
Effects of selected CAM therapies on duration of pain change. | 5 hours
  We will examine the effectiveness of CAM therapies on repeated measures of self-reported pain over several hours after therapy to assess the distribution and decay of the pain change effect.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Dusek, PhD, Principal Investigator — Allina Health
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Dusek JA, Rivard RL, Griffin KH, Finch MD. Significant Pain Reduction in Hospitalized Patients Receiving Integrative Medicine Interventions by Clinical Population and Accounting for Pain Medication. J Altern Complement Med. 2021 Mar;27(S1):S28-S36. doi: 10.1089/acm.2021.0051. PMID 33788611